CLINICAL TRIAL: NCT05926635
Title: Efficacy of a Rehabilitation Program With the Pediatric Exoskeleton ATLAS 2030 in Pediatric Patients With Cerebral Palsy
Status: Active, not recruiting | Type: Observational
Sponsor: MarsiBionics (Industry)
Collaborators: National Research Council, Spain (Other Government); Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); Hospital Universitario La Paz (Other); Hospital Universitario 12 de Octubre (Other); Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Other Study IDs: SERMAS
Record Dates: First submitted 2023-05-23; First posted 2023-07-03 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy
Keywords: exoskeleton; cerebral palsy; gait; rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exoskeleton group: sessions of rehabilitation with the ATLAS 2030 exoskeleton twice per week as part of their of their routine rehabilitation
  Interventions: Device: ATLAS 2030
- Control group: The children included in the control group will continue receiving their usual conventional therapy

INTERVENTIONS:
Device: ATLAS 2030 — sessions of rehabilitation with the ATLAS 2030 exoskeleton twice per week as part of their routine rehabilitation
  Groups: Exoskeleton group

SUMMARY:
Cerebral Palsy (CP) is the first cause of motor disability in children worldwide. ATLAS 2030 is a robotic gait exoskeleton designed to rehabilitate children with motor disability. The objective of this study is to analyse the efficacy of a training program with ATLAS 2023 in chilren with CP.

DETAILED DESCRIPTION:
A sample of children with CP will be divided into 2 groups, the experimental group will receive 32 sesions withe the ATLAS 2030 exoskeleton, whereas the control group will continue to receive their regular conventional therapy. Assessments will be performed at the beginning and the end of the intervention, as well as after 6, 9 and 12 months of the end of the intervention for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Medical authorization for standing, gait training and weight bearing.
* Informed consent signed by legal guardians.
* Confirmed diagnosis of cerebral palsy GMFCS levels III or IV.
* Proper family acceptance and commitment level.
* Receiving a minimum of 2 hours of therapy/activities promoting physical activity.
* Maximum user weight of 35 kg.
* Hip width (between greater trochanteres) less than or equal to 35 cm.
* Length of the thigh (distance from the greater trochanter to the lateral condyle of the tibia) from 24cm to 33cm.
* Tibia leg length (distance from the lateral condyle of the tibia to the lateral malleolus) from 23cm to 32cm.
* Shoe size 27-33 (EU)

Exclusion Criteria:

* More than 8 sessions of robotic therapy during a month in the previous year to the beginning of the study.
* Intensive rehabilitation during the study.
* Imposibility of the family to fulfill treatment calendar.
* Spasticity equal to 4 on the Modified Ashworth Scale at the time of use of the device.
* More than 20º of hip and/or knee flessum at the time of using the exoskeleton.
* Necessity to walk with 10º of hip abduction.
* Necessity to walk with more than 9º of ankle dorsiflexion or plantar flexion or impossibility to use an orthosis to reach 90º in the ankle joint.
* Severe skin lesion on parts of the lower extremities that are in contact with the device.
* Scheduled surgery (rachis, limbs) for the duration of the study or surgery performed (rachis, extremities) in the last 6 months.
* History of fracture without trauma. History of bone fracture traumatic in lower extremities or pelvic girdle in the last 3 months.
* Severe rigid orthopedic deformities of the spine and/or lower limbs.
* Cognitive or conductual disorders that may lead to a lack of adherence to the attachment to the device.
* Conditions that provoke exercise intolerance.
* Conductual disorders that may interfere with the use of the device or their participation in the study, like impulsiveness or the inability to understand simple comands.
* Allergy to any of the ATLAS materials: cotton, nylon, polyester, polyamide, polyethylene or propylene.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with cerebral palsy with Gross Motor Function Classification level III (children walk using a hand-held mobility device in most indoor settings) or IV (children use methods of mobility that require physical assistance or powered mobility in most settings).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-05-11 (Estimated); Study Completion 2025-05-11 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure-88 (GMFM-88) | At the beginning and the end of the intervention (4 months), as well as after 6, 9 and 12 months (follow-up)
  To measure changes in gross motor function in children with cerebral palsy using the Gross Motor Functional Measure-88.
  The minimum value is 0 and the maximum value is 100 .When the GMFM score is lower, the skill level is lower.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Through study completion, along 1 year
  changes in spasticity measured by the Modified Ashworth Scale (MAS). The spasticity of each muscle group is measured with a scale scored from 0 to 4, where 0 means no spasticity and 4 means the joint is fixed and therefore, the highest level of spasticity
Pediatric Quality of Life Inventory (PedsQLTM) | At the beginning and the end of the intervention (4 months), as well as after 6, 9 and 12 months (follow-up)
  Changes in self perceived quality of life measured by the Pediatric Quality of Life Inventory (PedsQLTM). Every item is measured on a scale from 0 (higher quality of life) to 4 (lower quality of life)
Changes in Gait Deviation Index (GDI) | At the beginning and the end of the intervention (4 months), as well as after 6, 9 and 12 months (follow-up)
  Changes in Gait Deviation Index (GDI) measured with a tridimensional motion analysis system

CONTACTS AND LOCATIONS:
Overall Officials: Olga Arroyo Riaño, Principal Investigator — Hospital Universitario Gregorio Marañón; María Teresa Vara Arias, Principal Investigator — Hospital Infantil Universitario Niño Jesús; Ignacio Martínez Caballero, Principal Investigator — Hospital Infantil Universitario Niño Jesús; Sandra Espinosa García, Principal Investigator — Hospital Univsersitario La Paz; Sofía García de las Peñas, Principal Investigator — Hospital 12 de Octubre; Elena García Armada, Principal Investigator — National Research Council, Spain
Locations (5):
- Spain (5):
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Infantil Universitario Niño Jesús-Servicio de Rehabilitación, Madrid
  - Hospital Universitario Niño Jesús-Servicio de Neuro Ortopedia, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No